CLINICAL TRIAL: NCT03984799
Title: Interleukin-5 Receptor Expression in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Larry Borish, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21547
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchoscopy (Experimental): Research bronchoscopy
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Samples obtained during bronchoscopy and blood samples will be evaluated to define inflammatory markers of COPD
  Other Names: Blood Draw

SUMMARY:
At visit one, after the subject has signed the consent form, subjects will answer questions and have maximum reversibility lung function test to determine if they are eligible to proceed with the study. Once the study team has proven that the subject is eligible to proceed the study team will collect a sputum sample and blood sample to study their cells. At visit two the subjects will undergo a research bronchoscopy at this point the study team will collect more samples including a BAL sample and another blood sample. Three follow up phone calls will be conducted after the procedure to ensure subject safety, the study team will record any symptoms that they are experiencing at that time. Throughout this study the samples will be analyzed to see if a larger subset of COPD patients could benefit from using the drug mepolizumab.

DETAILED DESCRIPTION:
During this study the subjects will have a bronchoscopy where the study team will collect airway samples to see how the subjects express certain cells. The subjects will also have two blood draws to provide information on the number of inflammatory cells that are present in their blood. This will help the study team determine if mepolizumab might be able to be used in more patients with COPD. The use of mepolizumab in COPD subjects with elevated blood eosinophils has been proven effective. However, the cellular mechanisms in the COPD population are unknown, including the extent to which these subjects express IL-5 in their airway and whether eosinophils are the sole target. Through this study the study team plans to provide proof of concept that mepolizumab could target additional IL-5-expressing immune cells in the airway, including especially PMNs. The study team will also investigate additional feasible biomarkers that could be utilized to predict mepolizumab responsiveness in COPD. The study team is hoping to determine if COPD patients with elevated blood eosinophils will demonstrate increased concentrations of IL-5 in their bronchoalveolar lavage (BAL) fluid and increased expression in their BAL of CD125+ PMNs. To address this hypothesis, the following specific aims will be addressed: To define the expression of IL-5R on PMNs in COPD and to demonstrate elevated concentrations of IL-5 in BALF obtained from COPD subjects with blood eosinophils (≥300/µL).

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥40 and ≤80.

  * COPD according to ATS-ERS guidelines
  * Current or former smokers (≥10 pack-years) / non-smokers without a history of asthma
  * FEV1/FVC ratio 0.70 before and after bronchodilator
  * FEV1 after bronchodilator ≥50% predicted and <80% predicted
  * No recent exacerbation within 30 days of bronchoscopy
  * No symptoms of recent symptomatic infection (change in sputum volume or color in the previous 30 days).
  * Absolute eosinophil count >300/µL within one month of the research bronchoscopy.

Exclusion Criteria:

* • Current diagnosis of asthma

  * Non-smokers with a history of asthma
  * Recent exacerbation within 30 days of bronchoscopy
  * Major medical co-morbid or primary disorder including systemic disorders involving the heart, CNS, renal, and endocrine systems
  * Positive pregnancy test at time of bronchoscopy in women of child-bearing years
  * Recent change in COPD control regimen (within 60 days). Stable orally-dosed CCS will not be a contraindication to study as long as the dose was not changed within 60 days.
  * Recent (with 1-year) administration of a biologic agent
  * Presence of allergic sensitization (atopy) (if obtained) will not be considered an exclusion.
  * Presence of hypereosinophil syndrome (HES), eosinophilic granulomatous polyangiitis (EGPA), nasal polyposis, helminth infection, or any other medical condition associated with eosinophilia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
IL-5R expression on bronchial neutrophils | within 24 hours
  IL-5R will be quantified on neutrophils purified from bronchoalveolar lavage fluid
IL-5 concentration in BALF | within 24 hours
  IL-5 will be quantified in bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borish L, Teague WG, Patrie JT, Wavell KW, Barros AJ, Malpass HC, Lawrence MG. Further evidence of a type 2 inflammatory signature in chronic obstructive pulmonary disease or emphysema. Ann Allergy Asthma Immunol. 2023 May;130(5):617-621.e1. doi: 10.1016/j.anai.2023.01.024. Epub 2023 Feb 2. PMID 36736724